CLINICAL TRIAL: NCT04533932
Title: Endosonographic Real-time and Shear Wave Elastography to Assess Liver stiffness-a Pilot Study
Brief Title: Endosonographic Shear Wave Elastography for Liver Stiffness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Olympus Corporation of the Americas (Industry)
Responsible Party: Principal Investigator, Divyanshoo Kohli, MD, Director of Endoscopy, Kansas City Veteran Affairs Medical Center
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: MBRF
Record Dates: First submitted 2020-08-23; First posted 2020-09-01 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elastography
  Interventions: Diagnostic Test: Elastography

INTERVENTIONS:
Diagnostic Test: Elastography — Endosonographic shear wave elastography

SUMMARY:
This is a single-center, prospective, non-randomized, comparative study which will compare the diagnostic accuracy and safety of endosonographic real-time Elastography and shear wave Elastography with the current standards of care, i.e. liver biopsy and Vibration-controlled transient elastography (Fibroscan). Subjects who are referred for an endoscopic ultrasound (EUS) guided liver biopsy will be prospectively enrolled to undergo liver biopsy, Elastography and/or Vibration-controlled transient elastography.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for EUS guided liver biopsy
* Elevated liver enzymes without obvious etiology, thus necessitating liver biopsy or clinical concern for cirrhosis or NASH requiring histological confirmation
* Ability to provide informed consent and willing to participate

Exclusion Criteria:

* Clinical evidence of cirrhosis which obviates need for liver biopsy
* Noninvasive lab testing which confirms presence of cirrhosis
* Surgically altered foregut anatomy which precludes safe endoscopic liver biopsy
* Coagulopathy with INR greater than 1.6 in patients on anticoagulant therapy
* Thrombocytopenia with platelet count less than 50,000/mL
* Pregnancy (positive urine pregnancy test in females of childbearing age)
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver biopsy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Degree of fibrosis | through study completion, an average of 1 year
  Degree of fibrosis based on histological assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Kohli DR, Mettman D, Andraws N, Haer E, Porter J, Ulusurac O, Ullery S, Desai M, Siddiqui MS, Sharma P. Comparative accuracy of endosonographic shear wave elastography and transcutaneous liver stiffness measurement: a pilot study. Gastrointest Endosc. 2023 Jan;97(1):35-41.e1. doi: 10.1016/j.gie.2022.08.035. Epub 2022 Aug 29. PMID 36049537